CLINICAL TRIAL: NCT01514981
Title: A Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of AMG 761 in Subjects With Asthma
Brief Title: AMG 761 in Adults With Asthma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Administrative decision
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Basic Science
Other Study IDs: 20080451
Record Dates: First submitted 2011-12-19; First posted 2012-01-23 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-04

CONDITIONS: Asthma
Keywords: Asthma
MeSH Terms: conditions — Asthma | interventions — mogamulizumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- AMG 761 (Experimental)
  Interventions: Drug: AMG 761
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AMG 761 — Single dose of AMG 761 on study day 1.
  Arms: AMG 761
Drug: Placebo — Single dose of placebo on study day 1.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine that no significant safety issues will be identified following a single dose of AMG 761 in asthma subjects that would preclude further development of AMG 761.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, with no history or evidence of clinically relevant medical or psychiatric disorders (with the exception of asthma) as determined by the investigator in consultation with the Amgen physician where medically appropriate
* Immunizations up to date, with a minimum of tetanus, diphtheria, pertussis (td/Tdap), pneumococcal (polysaccharide), influenza (during flu season) and H1N1 (where and when available) vaccinations, as determined by the principal investigator
* Body mass index (BMI) in the range of 18 to 35 kg/m2, inclusive
* Is a current non-smoker and has not used any tobacco products within the last 6 months and the cumulative smoking history must be ≤ 10 pack years
* Clinically stable with a physician diagnosis of asthma for a minimum of 6 months prior to enrollment, and with no change in asthma treatment for at least 3 months prior to enrollment. As needed beta-agonist use (ie, PRN) should be considered a stable treatment
* Documented history of atopy to oak, mite, ragweed, timothy grass, Alternaria mold, kochia pollen, aspergillus, or cottonwood within 18 months or positive atopy skin prick test for these specific allergens during the screening period
* Additional inclusion criteria apply

Exclusion Criteria:

* Past history of serious skin rash requiring hospitalization
* Active, or history of (within 12 months of enrollment), acute viral infection of the skin (eg, herpes simplex, herpes zoster, or molluscum contagiosum)
* Active or history of psoriasis, or a first degree relative with active or known history of psoriasis
* First degree relatives with active or history of systemic lupus erythematosus or type 1 diabetes, rheumatoid arthritis or other active autoimmune disorder, as determined by the principal investigator
* History of life-threatening anaphylaxis
* Experienced an asthma exacerbation (defined as a disease episode resulting in treatment in an emergency room, hospitalization, or an episode treated with oral corticosteroids in dosage of at least 5 mg/day prednisone or equivalent for ≥ 1 week) during the 6 months prior to enrollment
* Additional exclusion criteria apply

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2011-12; Primary Completion 2014-01 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
The number of treatment emergent adverse events per subject including clinically significant changes in vital signs, physical examinations, laboratory safety tests and ECGs. | 16 weeks
The number of subjects with anti-AMG 761 antibodies after a single dose of AMG 761. | 16 weeks

SECONDARY OUTCOMES:
The maximum observed concentration, time to maximum concentration and the area under the serum concentration-time curve after a single dose of AMG 761. | 16 weeks
The circulating CD4+ CCR4+ T cell count. | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (2):
- United States (2):
  - Research Site, Denver, Colorado
  - Research Site, Miami, Florida

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com